CLINICAL TRIAL: NCT02154438
Title: The Effect of Ketamine Infusion for Reduction of Neuropathic Pain and Improvement of Quality of Life After Lumbar Surgery
Brief Title: The Effect of Ketamine Infusion on Lumbar Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Cholhee Park, Clinical assistant professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-2014-0062
Record Dates: First submitted 2014-05-25; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketamine (Experimental): ketamine 0.5mg/kg loading dose and followed by 0.5mg/kg/h during operation
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): normal saline 0.5mg/kg loading dose and followed by 0.5mg/kg/h during operation

INTERVENTIONS:
Drug: Ketamine — ketamine 0.5mg/kg loading followed by 0.5mg/kg/h infusion during operation
  Other Names: Huons ketamine hch injection
  Arms: ketamine

SUMMARY:
The purpose of this study is to evaluate the effect of ketamine infusion for reduction of neuropathic pain and improvement of quality of life after lumbar surgery.

DETAILED DESCRIPTION:
Neuropathic pain defined as 'pain caused by a lesion or disease of the somatosensory system'. Neuropathic pain is 20 - 35% of low back pain.

Ketamine is categorized as N-methyl D-aspartate receptor antagonist. Ketamine has an analgesic effect in low dose and anesthetic effect in relative high dose. Also, ketamine is used in chronic neuropathic pain as postherpetic neuralgia., phantom pain, central neuropathic pain, complex regional pain syndrome, ischemic pain.

In this study, ketamine will be infused during lumbar surgery in randomized, double-blind and double-blind parallel group control trial.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing lumbar spine surgery due to back pain patients
* American Physical Status Classification I or II

Exclusion Criteria:

* less than 3 month of back pain
* past history of operation at lumbar area
* past history of glucoma, drug abuse, alcohol abuse
* pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 1 day before lumbar surgery
  VAS score in 1 day before lumbar surgery
Pain Scores on the Visual Analog Scale | 1 month after lumbar surgery
  VAS score in 1 month after lumbar surgery
Pain Scores on the Visual Analog Scale | 3 month after lumbar surgery
  VAS score in 3 month after lumbar surgery

SECONDARY OUTCOMES:
Leeds assessment of neuropathic symptoms and signs (LANSS) score | 1 day before lumbar surgery
  LANSS score in 1 day before lumbar surgery
Leeds assessment of neuropathic symptoms and signs (LANSS) score | 1 month after lumbar surgery
  LANSS score in 1 month after lumbar surgery
Leeds assessment of neuropathic symptoms and signs (LANSS) score | 3 month after lumbar surgery
  LANSS score in 3 month after lumbar surgery
neuropathic pain scale (NPS) score | 1 day before lumbar surgery
  NPS score in 1 day before lumbar surgery
neuropathic pain scale (NPS) score | 1 month after lumbar surgery
  NPS score in 1 month after lumbar surgery
neuropathic pain scale (NPS) score | 3 month after lumbar surgery
  NPS score in 3 month after lumbar surgery
Oswestry disability index (ODI) score | 1 day before lumbar surgery
  ODI score in 1 day before lumbar surgery
Oswestry disability index (ODI) score | 1 month after lumbar surgery
  ODI score in 1 month after lumbar surgery
Oswestry disability index (ODI) score | 3 month after lumbar surgery
  ODI score in 3 month after lumbar surgery
WHO Quality of Life (WHOQOL-BREF) score | 1 day before lumbar surgery
  WHOQOL-BREF score in 1 day before lumbar surgery
WHO Quality of Life (WHOQOL-BREF) score | 1 month after lumbar surgery
  WHOQOL-BREF score in 1 month after lumbar surgery
WHO Quality of Life (WHOQOL-BREF) score | 3 month after lumbar surgery
  WHO Quality of Life (WHOQOL-BREF) score in 3 month after lumbar surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hyun Kim, MD, Principal Investigator — Department of Neurosurgery, The Spine and Spinal Cord Institute, Gangnam Severance Spine Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea